CLINICAL TRIAL: NCT02922829
Title: The PreNAPS Study: Food Insecurity, Prenatal Nutrition, and Psychosocial Health Outcomes Among HIV Infected and Uninfected Pregnant Women Attending ANC Services at Gulu Regional Referral Hospital
Brief Title: The PreNAPS Study: FI, Nutrition, and Psychosocial Health Outcomes at Gulu Regional Referral Hospital
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Cornell University (Other); Tufts University (Other); Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: 1206003141
Record Dates: First submitted 2016-09-26; First posted 2016-10-04 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: HIV; Pregnancy
Keywords: Food Insecurity; Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Prenatal Nutrition and Psychosocial Health Outcomes (PreNAPS) study was a two year collaboration between Gulu, Makarere, Cornell, and Tufts Universities. The PreNAPs study's primary goals were: a) to determine the differential impacts of food insecurity on gestational weight gain and prenatal depression, and b) to elucidate the mechanisms underlying the relationship between food insecurity and weight gain and/depression among HIV infected and HIV uninfected pregnant women in Gulu, Northern Uganda.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Known HIV status
* Receiving antiretroviral therapy (if HIV-infected)
* Attending antenatal care at Gulu Regional Referral Hospital
* >18 years of age

Exclusion Criteria:

* Pregnant women <18 years of age
* Unknown HIV status
* Not receiving antiretroviral therapy (if HIV-infected)
* Not attending antenatal care at Gulu Regional Referral Hospital

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women were enrolled during pregnancy at Gulu Regional Referral Hospital antenatal clinic in Gulu, Uganda
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Impacts of food insecurity (IFIAS) on gestational weight gain (kg) among pregnant women of mixed HIV status in Gulu, Uganda | Approximately 1 year
  Explore the underlying mechanisms and impacts of food insecurity (using the Individuals Food Insecurity Access Scale (IFIAS)) on gestational weight gain (kg) among pregnant women of mixed HIV status in Gulu, Uganda.

SECONDARY OUTCOMES:
Impacts of food insecurity on maternal depression among pregnant women of mixed HIV status in Gulu, Uganda. | Approximately 1 year
  Explore the underlying mechanisms and impacts of food insecurity on maternal depressive symptoms among pregnant women of mixed HIV status in Gulu, Uganda.

CONTACTS AND LOCATIONS:
Overall Officials: Sera L Young, MA, PhD, Principal Investigator — Northwestern University; Barnabas K Natamba, MPH, PhD, Principal Investigator — Michigan State University
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Natamba BK, Mehta S, Achan J, Stoltzfus RJ, Griffiths JK, Young SL. The association between food insecurity and depressive symptoms severity among pregnant women differs by social support category: a cross-sectional study. Matern Child Nutr. 2017 Jul;13(3):e12351. doi: 10.1111/mcn.12351. Epub 2016 Aug 9. PMID 27507230
- [Background] Natamba BK, Kilama H, Arbach A, Achan J, Griffiths JK, Young SL. Reliability and validity of an individually focused food insecurity access scale for assessing inadequate access to food among pregnant Ugandan women of mixed HIV status. Public Health Nutr. 2015 Nov;18(16):2895-905. doi: 10.1017/S1368980014001669. Epub 2014 Aug 29. PMID 25171462
- [Background] Natamba BK, Achan J, Arbach A, Oyok TO, Ghosh S, Mehta S, Stoltzfus RJ, Griffiths JK, Young SL. Reliability and validity of the center for epidemiologic studies-depression scale in screening for depression among HIV-infected and -uninfected pregnant women attending antenatal services in northern Uganda: a cross-sectional study. BMC Psychiatry. 2014 Nov 22;14:303. doi: 10.1186/s12888-014-0303-y. PMID 25416286
- [Derived] Lane CE, Widen EM, Collins SM, Young SL. HIV-Exposed, Uninfected Infants in Uganda Experience Poorer Growth and Body Composition Trajectories than HIV-Unexposed Infants. J Acquir Immune Defic Syndr. 2020 Oct 1;85(2):138-147. doi: 10.1097/QAI.0000000000002428. PMID 32604132
- [Derived] Widen EM, Collins SM, Khan H, Biribawa C, Acidri D, Achoko W, Achola H, Ghosh S, Griffiths JK, Young SL. Food insecurity, but not HIV-infection status, is associated with adverse changes in body composition during lactation in Ugandan women of mixed HIV status. Am J Clin Nutr. 2017 Feb;105(2):361-368. doi: 10.3945/ajcn.116.142513. Epub 2017 Jan 4. PMID 28052888